CLINICAL TRIAL: NCT03434288
Title: Pilot Evaluation of PCR Multiplex Tests for a Rapid Diagnosis of Bone Infections in Diabetic Foot
Brief Title: Assessment of PCR Multiplex Tests as a Tool to Obtain a Quicker Diagnosis of Bacteria Responsible for Foot Osteomyelitis Than Usual Cultures
Acronym: RAPDIAGOS
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0013
Record Dates: First submitted 2018-01-26; First posted 2018-02-15 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Diabetes Mellitus; Foot Osteomyelitis
Keywords: Diabetes; Diabetic foot; Osteomyelitis
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot; Osteomyelitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetic patients with foot osteomyelitis: Biological and MRI signs of foot osteomyelitis
  Interventions: Other: Bone sampling

INTERVENTIONS:
Other: Bone sampling — Bone biopsy in Diabetic patients with foot osteomyelitis

SUMMARY:
Bone samples from infected diabetic feet will be collected and tests will be performed for the diagnosis of causative bacteria. Samples will be processed by PCR multiplex tests and usual cultures for identification of causative bacteria and sensitivity to antibiotics. Results obtained by the two methods will be compared in terms of quickness and similarity of germ identification. Usual care strategy will not be modified since results of PCR multiplex tests will not be transmitted to the physicians before the results of usual cultures.

DETAILED DESCRIPTION:
This study will investigate the quickness of identification of bacteria causing bone infection in the feet of patients with diabetes from bone samples obtained by biopsies performed in usaual care practice.

Bone biopsies will be performed in patients diagnosed for osteomyelitis from clinical, biological and MRI signs. Bone samples will be collected in Ultra-Turrax® tubes in the operating theater before being transferred to the department of bacteriology. Time of registration at the bacteriology lab will be considered as Time 0 (T0).

Samples will be processed simultaneously using the usual culture method and by PCR Multiplex tests.

The time of identification of causative bacteria for bone infection (time 1, T1) and the time of identification of sensitivity/resistance to antibiotics (time 2, T2) by the two different methods will be recorded.

Identified germs and their sensitivity/resistance to antibiotics according to the two methods will be compared.

If the results are similar, the time that could be gained for the prescription of specific antibiotics from PCR multiplex tests' results will be computed in comparison to the prescription performed from the results of usual cultures.

ELIGIBILITY:
Inclusion criteria:

* Biological and MRI signs of foot osteomyelitis
* Indication of bone biopsy
* No antibiotics since 2 weeks

Exclusion criteria:

* Antibiotic therapy
* Previous cultures for the same infectious event

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients admitted in hospital for foot osteomyelitis
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Time for identification of bacteria responsible for foot osteomyelitis | 12-48 hours
  The difference of time between usual cultures and PCR multiplex tests to identify responsible bacteria will be assessed

SECONDARY OUTCOMES:
Time for identification of sensitivity/resistance to antibiotics of the bacteria responsible for foot osteomyelitis | 12-96 hours
  The difference of time between usual cultures and PCR multiplex tests to identify sensitivity/resistance to antibiotics of responsible bacteria for foot osteomyelitis will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Eric RENARD, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC